CLINICAL TRIAL: NCT06342596
Title: A Phase 1, Open-Label, Two-Part Study of the Disposition and Absolute Bioavailability of [14C]-LY3473329 in Healthy Male Participants
Brief Title: A Study of Carbon-14-Labelled [14C] LY3473329 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 18597; J2O-MC-EKBD (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-02-26; First posted 2024-04-02 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Healthy
Keywords: Radioactive; ADME; Disposition; Bioavailability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- [14C]-LY3473329 (Part 1) (Experimental): Single dose of [¹⁴C]-LY3473329 administered orally
  Interventions: Drug: [14C]-LY3473329
- LY3473329 + [14C]-LY3473329 (Part 2) (Experimental): Single dose of LY3473329 administered orally followed by a single dose of [¹⁴C]-LY3473329 administered intravenously (IV)
  Interventions: Drug: [14C]-LY3473329; Drug: LY3473329

INTERVENTIONS:
Drug: [14C]-LY3473329 — Administered orally
  Arms: [14C]-LY3473329 (Part 1)
Drug: [14C]-LY3473329 — Administered IV
  Arms: LY3473329 + [14C]-LY3473329 (Part 2)
Drug: LY3473329 — Administered orally
  Arms: LY3473329 + [14C]-LY3473329 (Part 2)

SUMMARY:
The main purpose of this study is to evaluate how much of the study drug (LY3473329), administered as a single dose that has the radioactive substance 14C incorporated into it, passes from blood into urine, feces and expired air in healthy male participants. The study will also measure how much of the study drug gets into the bloodstream when taken orally, compared to when injected directly into the vein, how its broken down, and how long it takes the body to get rid of it. The study is conducted in two parts. The study will last up to approximately 9 and 7 weeks for part 1 and 2, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Male participants who are overtly healthy as determined by medical evaluation
* Have a body mass index of 18.0 to 35.0 kilograms per meter squared (kg/m²), inclusive
* Males who agree to use highly effective or effective methods of contraception

Exclusion Criteria:

* Have known allergies to LY3473329, related compounds, or any components of the formulation, or history of significant atopy
* Have a history of constipation or have had acute constipation within 3 weeks prior to check-in
* Have participated in any clinical study involving a radiolabeled investigational product within 12 months prior to check-in. Any previous radiolabeled study intervention must have been received more than 12 months prior to check-in
* Have used or plan to use over-the-counter or prescription medication within 14 days prior to dosing, or any medications or products known to alter drug absorption, metabolism, or elimination processes
* Have participated, within the last 3 months, in a clinical study involving an investigational product

Ages: 35 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 16 (Actual)
Dates: Start 2024-03-05 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Part 1: Urinary Excretion of LY3473329 Radioactivity Over Time Expressed as a Percentage of the Total Radioactive Dose Administered | Day 1 up to Day 29 post dose
  Part 1: Urinary Excretion of LY3473329 Radioactivity Over Time Expressed as a Percentage of the Total Radioactive Dose Administered
Part 1: Fecal Excretion of LY3473329 Radioactivity Over Time Expressed as a Percentage of the Total Radioactive Dose Administered | Day 1 up to Day 29 post dose
  Part 1: Fecal Excretion of LY3473329 Radioactivity Over Time Expressed as a Percentage of the Total Radioactive Dose Administered
Part 2: Pharmacokinetics (PK): Absolute bioavailability (F) of LY3473329 | Day 1 up to Day 9 post dose
  Part 2: PK: F of LY3473329

SECONDARY OUTCOMES:
Part 1: PK: Area Under the Curve Concentration Versus Time Curve From Time zero to Last Time Point (AUC[0-tlast]) of LY3473329 | Day 1 up to Day 29 post dose
  Part 1: PK: AUC(0-tlast) of LY3473329
Part 1: PK: Area Under the Curve Concentration Versus Time Curve From Time zero to Last Time Point (AUC[0-tlast]) of Total Radioactivity | Day 1 up to Day 29 post dose
  Part 1: PK: AUC(0-tlast) of Total Radioactivity
Part 1: PK: Area Under the Curve Concentration Versus Time Curve From Time zero to Infinity (AUC[0-∞) of LY3473329 | Day 1 up to Day 29 post dose
  Part 1: PK: AUC(0-∞) of LY3473329
Part 1: PK: Area Under the Curve Concentration Versus Time Curve From Time zero to Infinity (AUC[0-∞) of Total Radioactivity | Day 1 up to Day 29 post dose
  Part 1: PK: AUC(0-∞) of Total Radioactivity
Part 1: PK: Maximum Concentration (Cmax) of LY3473329 | Day 1 up to Day 29 post dose
  Part 1: PK: Cmax of LY3473329
Part 1: PK: Maximum Concentration (Cmax) of Total Radioactivity | Day 1 up to Day 29 post dose
  Part 1: PK: Cmax of Total Radioactivity
Part 1: Total Radioactivity Recovered in Urine, Feces, and Expired Air (if applicable) | Day 1 up to Day 29 post dose
  Part 1: Total Radioactivity Recovered in Urine, Feces, and Expired Air (if applicable)
Part 1: Total Number of Metabolites of LY3473329 | Day 1 up to Day 29 post dose
  Part 1: Total Number of Metabolites of LY3473329
Part 2: PK: AUC (0-∞) of LY3473329 | Day 1 up to Day 9 post dose
  Part 2: PK: AUC (0-∞) of LY3473329
Part 2: PK: AUC (0-∞) of [14C]-LY3473329 | Day 1 up to Day 9 post dose
  Part 2: PK: AUC (0-∞) of [14C]-LY3473329
Part 2: PK: AUC (0-∞) of Total Radioactivity | Day 1 up to Day 9 post dose
  Part 2: PK: AUC (0-∞) of Total Radioactivity
Part 2: PK: Cmax of LY3473329 | Day 1 up to Day 9 post dose
  Part 2: PK: Cmax of LY3473329
Part 2: PK: Cmax of [14C]-LY3473329 | Day 1 up to Day 9 post dose
  Part 2: PK: Cmax of [14C]-LY3473329
Part 2: PK: Cmax of Total Radioactivity | Day 1 up to Day 9 post dose
  Part 2: PK: Cmax of Total Radioactivity
Part 2: Total Radioactivity Recovered in Urine and Feces | Day 1 up to Day 9 post dose
  Part 2: Total Radioactivity Recovered in Urine and Feces

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Fortrea Clinical Research Unit, Holbeck, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No